CLINICAL TRIAL: NCT04846634
Title: Penpulimab-based Combination Neoadjuvant/Adjuvant Therapy for Patients With Resectable Locally Advanced Non-small Cell Lung Cancer: a Phase II Clinical Study (ALTER-L043)
Acronym: ALTER-L043
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Collaborators: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ALTER-L043
Record Dates: First submitted 2021-04-14; First posted 2021-04-15 (Actual); Last update posted 2021-04-15 (Actual); Status verified 2021-04

CONDITIONS: Resectable Locally Advanced Non-small Cell Lung Cancer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- neoadjuvant Penpulimab + chemotherapy followed by adjuvant Penpulimab (Experimental)
  Interventions: Drug: Penpulimab+Cisplatin/Carboplatin+Pemetrexed/Paclitaxel/Gemcitabine/Docetaxel
- neoadjuvant Penpulimab + chemotherapy + Anlotinib followed by adjuvant Penpulimab + Anlotinib. (Experimental)
  Interventions: Drug: Penpulimab+Anlotinib+Cisplatin/Carboplatin+Pemetrexed/Paclitaxel/Gemcitabine/Docetaxel
- neoadjuvant Penpulimab + Anlotinib followed by adjuvant Penpulimab + Anlotinib. (Experimental)
  Interventions: Drug: Penpulimab+Anlotinib

INTERVENTIONS:
Drug: Penpulimab+Cisplatin/Carboplatin+Pemetrexed/Paclitaxel/Gemcitabine/Docetaxel — A cycle of treatment is defined as 21 days of once daily treatment.
  Other Names: Investigational Product
  Arms: neoadjuvant Penpulimab + chemotherapy followed by adjuvant Penpulimab
Drug: Penpulimab+Anlotinib+Cisplatin/Carboplatin+Pemetrexed/Paclitaxel/Gemcitabine/Docetaxel — A cycle of treatment is defined as 21 days of once daily treatment.
  Other Names: Investigational Product
  Arms: neoadjuvant Penpulimab + chemotherapy + Anlotinib followed by adjuvant Penpulimab + Anlotinib.
Drug: Penpulimab+Anlotinib — A cycle of treatment is defined as 21 days of once daily treatment.
  Other Names: Investigational Product
  Arms: neoadjuvant Penpulimab + Anlotinib followed by adjuvant Penpulimab + Anlotinib.

SUMMARY:
This is a multicenter, randomized, open label, phase II study.

DETAILED DESCRIPTION:
This is a multicenter, randomized, open label, phase II study assessing the efficacy and safety of penpulimab plus chemotherapy or penpulimab plus anlotinib or penpulimab plus chemotherapy and anlotinib as neoadjuvant/adjuvant treatment in patients with resectable locally advanced non-small cell lung cancer. Eligible patients will be randomized to receive either penpulimab (200mg, iv, Q3W) plus chemotherapy (platinum based chemotherapy) or penpulimab (200mg, iv, Q3W) plus anlotinib (12mg, po, day 1-14, Q3W) or penpulimab (200mg, iv, Q3W) plus chemotherapy (platinum based chemotherapy) and anlotinib (12mg, po, day 1-14, Q3W) in a 1:1:1 ratio.

ELIGIBILITY:
Inclusion Criteria:

* Early stage IIB-IIIB (N2), operable non-small cell lung cancer, confirmed in tissue.
* Epidermal growth factor receptor/anaplastic lymphoma kinase/ROS1 gene fusions mutation was negative in primary tumor or lymph node metastasis.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-1 with no deterioration over the previous 2 weeks and a minimum life expectancy of 12 weeks.
* Lung function capacity capable of tolerating the proposed lung surgery.
* Patients had never received surgery, chemotherapy, radiotherapy or biotherapy.

Exclusion Criteria:

* Large cell carcinoma and mixed cell lung cancer.
* Any systemic anti-cancer treatment for NSCLC, including cytotoxic drug therapy, immunotherapy, experimental treatment.
* Prior treatment with local radiotherapy.
* Prior treatment with any drug that targets T cell co-stimulations pathways (such as checkpoint inhibitors).
* Prior treatment with antilotinib and other antiangiogenic drugs.
* History of hypersensitivity to any active or inactive ingredient of Penpulimab, Anlotinib or chemotherapy.
* Patients with multiple factors affecting oral medication (e.g. inability to swallow, chronic diarrhea, and intestinal obstruction, etc.).
* Past medical history of interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonitis that required steroid treatment, or any evidence of clinically active interstitial lung disease.
* Patients whose tumor has invaded important blood vessels or whose tumor is likely to invade important blood vessels and cause fatal massive hemorrhage during follow-up study.
* Patients who have had arteriovenous thrombosis events within 6 months, such as cerebrovascular accident (including transient ischemic attack), deep venous thrombosis and pulmonary embolism.
* Pregnant or lactating women.
* History of neurological or mental disorders, including epilepsy or dementia.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-08 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Major pathological response (MPR) | About 3-6 weeks following completion of surgery.

SECONDARY OUTCOMES:
Objective response rate (ORR) | Within 7 days before surgery.
1 year Event-Free Survival rate | Up to 5 Years from randomization
Event-Free Survival (EFS) | Up to 5 years from randomization.
Overall survival (OS) | Up to 5 years from randomization.
Incidence of adverse events (AEs)/serious adverse events (SAEs) | Up to 5 Years from randomization

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi, China